CLINICAL TRIAL: NCT00627302
Title: Efficacy of PEG-400 and Systane Artificial Tears (Alcon) on Quality of Vision
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Eric Donnenfeld, MD, Ophthalmic Consultants of Long Island
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5353
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Myopia
Keywords: Quality of Vision
MeSH Terms: conditions — Myopia | interventions — polyethylene glycol 400

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 2 (Active Comparator): Systane
  Interventions: Drug: Systane
- 1 (Active Comparator): PEG-400
  Interventions: Drug: PEG-400

INTERVENTIONS:
Drug: PEG-400 — Day of Surgery: Starting 2 hours after surgery Instill one drop in randomized eye every two hours. Day 1-Week 1: Instill one drop in randomized eye four times daily
  Arms: 1
Drug: Systane — Day of Surgery: Starting 2 hours after surgery Instill one drop in randomized eye every two hours. Day 1-Week 1: Instill one drop in randomized eye four times daily
  Arms: 2

SUMMARY:
To evaluate the effect of PEG-400 and Systane on quality of vision after LASIK.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 21 years old
* Scheduled to undergo bilateral LASIK
* Likely to complete all study visits and able to provide informed consent

Exclusion Criteria:

* Prior or current use of topical cyclosporine within the last 1 year
* Known contraindications to any study medication or ingredients
* Ocular disorders
* Active ocular diseases or uncontrolled systemic disease
* Active ocular allergies
* Complications at the time of surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Quality of vision | 5 months

SECONDARY OUTCOMES:
Efficacy | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of long Island, Rockville Centre, New York, United States